CLINICAL TRIAL: NCT03065959
Title: A Phase 1b Study to Assess the Anti-fatigability Effect of CK-2127107 in Elderly Male and Female Subjects With Limitations in Mobility
Brief Title: A Study to Assess the Anti-fatigability Effect of CK-2127107 in Elderly Male and Female Subjects With Limitations in Mobility
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy determined at interim analysis
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Cytokinetics (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3318-CL-3001
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Mobility Limitation
Keywords: CK-2127107; Mobility Limitation; Phase 1b; skeletal muscle fatigue
MeSH Terms: conditions — Mobility Limitation | interventions — reldesemtiv

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CK-2127107, then Placebo (Experimental): Participants will first receive CK-2127107 tablets (twice daily) for 14 days. After a 14 day wash out period participants will then receive matching placebo.
  Interventions: Drug: reldesemtiv; Drug: Placebo
- Placebo, then CK-2127107 (Experimental): Participants will first receive Placebo tablets (twice daily) for 14 days. After a 14 day wash out period participants will then receive matching CK-2127107.
  Interventions: Drug: reldesemtiv; Drug: Placebo

INTERVENTIONS:
Drug: reldesemtiv — oral
  Other Names: CK-2127107
Drug: Placebo — oral

SUMMARY:
The purpose of this study is to investigate the effect of CK-2127107 versus placebo on skeletal muscle fatigue assessed as change from baseline versus 14 days of treatment in sum of peak torque during isokinetic knee extensions.

This study will also assess the effects of CK-2127107 on physical performance via a short physical performance battery (SPPB), stair-climb test and 6 minute walk test.

DETAILED DESCRIPTION:
Enrolled participants will be randomized to receive either CK-2127107 or Placebo first and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods of 14 days separated by a washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index of 18.5 to 35.0 kg/m2, inclusive.
* Subject has a score of greater than 4 and less than or equal to 10 on a Short physical performance battery (SPPB).
* Subject is able to complete the 6-minute walk test at screening without an assistive device or the help of another person.
* Subject is able to successfully complete the prestudy isokinetic knee extension (120 contractions). These assessments may be repeated once at the investigator's discretion (within the screening window).
* Subject is able to communicate well with the investigator and to understand and comply with the requirements of the study.
* Subject has a mini-mental state examination (MMSE) score of greater than 21 at screening.
* Subject is currently not following a a strenuous weekly exercise regimen.
* A sexually active male subject with female partner(s) of childbearing potential is eligible if:

  * Male subject agrees to use a male condom starting at screening and continue throughout study treatment and for 90 days after the final study drug administration.
  * If the male subject has not had a vasectomy or is not sterile as defined below, the male subject's female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continuing throughout study treatment and for 90 days after the male subject receives final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as from signing the informed consent form for the current study until completion of the Follow-up visit for this study.

Exclusion Criteria:

* Subject has had previous exposure to CK-2127107.
* Subject has any of the liver function tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, γ-glutamyl transferase and total bilirubin) above 1.5 times the upper limit of normal at day -1. In such a case, the assessment may be repeated once.
* Subject has an estimated glomerular filtration rate less than 30 mL/min per 1.73 m2 by the Cockcroft-Gault equation at screening.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding seasonal allergies) prior to study drug administration.
* Subject has/had a febrile illness or a symptomatic viral, bacterial (including upper respiratory infections), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has a serious cardiovascular disease, including a current New York Heart Association class II, class III or IV congestive heart failure or clinically significant valvular disease, history of cardiac arrest, uncontrolled angina or arrhythmia, chronic atrial fibrillation regardless of ventricular rate, persistent atrioventricular conduction block > first degree, or acute myocardial ischemic condition suspected on the Electrocardiogram (ECG) at screening (e.g., ST-segment elevation, down-sloping ST-segment depressions > 2 mm).
* Subject has myocardial infarction or other acute coronary syndrome, major heart surgery (i.e.,valve replacement or bypass surgery), stroke, deep vein thrombosis, or pulmonary embolus in the past 6 months prior to screening.
* Subject has any of the following, with or without blood pressure medication: a pulse < 40 or > 100 bpm; mean systolic blood pressure >160 mmHg; mean diastolic blood pressure > 100 mmHg (based on the measurements taken in triplicate after subject has been resting in seated position for 5 minutes; pulse will be measured automatically) at day 1. These assessments may be repeated once at the investigator's discretion (within the screening window).
* Subject has used the following drugs:

  * Strong cytochrome P450 (CYP) 3A4 inhibitor (e.g., itraconazole, clarithromycin; within 14 days prior to day 1
  * CYP3A4 inducer (e.g., barbiturates, rifampin) within 14 days prior to day 1.
  * Any medications known to affect physical function or muscle mass including androgen supplements, anti-androgens (such as luteinizing hormone-releasing hormone [LHRH] agonist, anti-estrogen [tamoxifen, etc],.), recombinant human growth hormone [rhGH] insulin, oral beta adrenergic agonists, megestrol acetate, dronabinol, metformin or other drugs) which might influence physical function or muscle mass within 6 weeks prior to screening.
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to screening.
* Subject has/had hemoglobin concentration below 10.0 g/dL at screening.
* Subject has/had > 20% weight loss in the previous 3 months prior to screening.
* Subject has/had chronic medications introduced within 2 weeks prior to screening.
* Subject has/had cancer requiring treatment currently or in the past 3 years (except primary nonmelanoma skin cancer, carcinoma in situ or cancers that have an excellent prognosis such as early stage breast or prostate cancer).
* Subject has/had a diagnosed neurological conditions or neuromuscular diseases causing impaired muscle function or mobility.
* Subject has current diagnosis of schizophrenia, other psychotic disorders or bipolar disorder.
* Subject has severe and/or uncontrolled medical conditions that could interfere with the study (e.g., severe neurological deficit after stroke, diabetic peripheral neuropathy, respiratory diseases requiring daytime supplemental oxygen, infection, gastrointestinal disorder, uncontrolled pain from osteoarthritis that would limit completion of study procedures or any other nonstable illness).
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibody, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, or antibodies to human immunodeficiency virus (HIV) type 1 at screening.
* Subject has/had a surgical procedure requiring general anesthesia within 2 months prior to screening, or a planned surgical procedure requiring general anesthesia during study period.
* Subject is using any nonmedical therapy, or dietary aids/food supplements that have not been at a stable dose for at least 4 weeks prior to baseline and/or are anticipated to change dosing regimen during the study.
* Subject has history of drug/chemical substance or alcohol abuse within 2 years prior to screening.
* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Change from period baseline in sum of the peak torque of 120 contractions | Baseline, Day 1 and Day 14 of Treatment Periods 1 and 2
  Peak torque measurements will be obtained with the participants seated and the knee extended through a determined range of motion. Peak torque (Nm) will be measured at 120°/second with 120 isokinetic contractions.

SECONDARY OUTCOMES:
Change from period baseline of Short physical performance battery (SPPB) score | Baseline, Day 1 and Day 14 of Treatment Periods 1 and 2
  Each of the 3 performance measures will be assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the test. A summary score (range 0-12) will be subsequently calculated by adding the 3 scores.
Change from period baseline of stair-climb test | Baseline, Day 1 and Day 14 of Treatment Periods 1 and 2
  Participants will be asked to ascend a set of 10 stairs. The participants will be asked to ascend the stairs 1 step at a time as quickly as the participant can while remaining safe. Time will be recorded as seconds.
Change from period baseline of distance walked assessed by 6-minute walk test | Baseline, Day 1 and Day 14 of Treatment Periods 1 and 2
  Participants will be instructed to walk as far as possible in 6 minutes, walking back and forth around the turn points. The distance will be recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Ohio University Heritage College, Athens, Ohio

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=378